CLINICAL TRIAL: NCT04374578
Title: Effect of Dulaglutide on Glycemic Variability in Patients With Type 2 Diabetes: A Multi-center Observational Study
Brief Title: Effect of Dulaglutide on Glycemic Variability in Patients With Type 2 Diabetes
Acronym: DIVE
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSE-202003
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dulaglutide 1.5 MG/ML — Dulaglutide 1.5Mg qw sc injection for 4 weeks

SUMMARY:
Glycemic variability will be assessed using continuous glucose monitor(CGM) in type 2 diabetic patients who receive dulaglutide 1.5 mg/qw injection for 4 weeks.

DETAILED DESCRIPTION:
Glycemic fluctuation is a major problem in glucose control in diabetic patients. It is interesting to know that whether weekly GLP-1RA can improve glycemic variability in diabetic patients. The present study aims to assess the effect of dulaglutide on glycemic variability using continuous glucose monitor(CGM) (Libra, Abbott) in type 2 diabetic patients with 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the test content and possible adverse reactions and voluntarily participate in the trial and sign the informed consent form;
* Meet the World Health Organization(WHO) (1999) criteria for the diagnosis and classification criteria for type 2 diabetes;
* 18 ≤ age ≤ 70 years old, male or female;

Exclusion Criteria:

* Subjects with Type 1 diabetes mellitus or secondary diabetes mellitus (i.e. any type other than T2DM)
* Personal history or family history of thyroid medullary carcinoma or multiple endocrine neoplasia type 2 (MEN2).
* History of pancreatitis or considered clinically at significant risk of developing pancreatitis during the course of the study (e.g. due to symptomatic gallstones).
* History of significant gastrointestinal (GI) surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function.
* Fasting triglyceride level more than 750 mg/dL at screening.
* Estimated Glomerular Filtration Rate (eGFR) less than 60 mL/minute/1.73 meter^2 (calculated using the Schwartz equation) at screening.
* ALT more than 2.5x upper limit of normal (ULN) or Bilirubin more than 1.5xULN (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin more than 35%) at screening.
* Use of a GLP-1receptor agonist at study entry and during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes come to the clinic who want to use dulaglutide and never used dulaglutide before
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Effect on glycemic variability | one months
  The FreeStyle Libre Pro (Abbott Co., Ltd) will be used to monitor glucose levels during the four weeks from the day before the first administration of the study drug

SECONDARY OUTCOMES:
Effect on Glycemic Control | one months
  It will be assessed at baseline and after one months of treatment to determine the anti-diabetic effect of dulaglutide

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No